CLINICAL TRIAL: NCT02711059
Title: Insulin Resistance in Primary Hyperparathyroidism, a Non-classical Manifestation
Brief Title: Insulin Resistance in Primary Hyperparathyroidism
Acronym: IRIPH
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: studien skjuts på framtiden
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Inga-Lena Nilsson, MD, PhD, consultant surgeon, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: KarolinskaUH_pHPT_diabetes
Record Dates: First submitted 2015-10-18; First posted 2016-03-17 (Estimated); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Hyperparathyroidism; Diabetes; Hypercalcemia
Keywords: hyperparathyroidism; insulin resistance
MeSH Terms: conditions — Hyperparathyroidism; Diabetes Mellitus; Hypercalcemia; Insulin Resistance | interventions — Parathyroidectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- parathyroidectomy (Active Comparator): change in insulin resistance
  Interventions: Procedure: parathyroidectomy
- control (No Intervention): the study participant will be examined parallel with the active comparator

INTERVENTIONS:
Procedure: parathyroidectomy — surgical treatment of hyperparathyroidism
  Other Names: parathyroid adenomectomy
  Arms: parathyroidectomy

SUMMARY:
The aims of this study is to analyse if insulin resistance in primary hyperparathyroidism (pHPT) is normalised after parathyroid adenomectomy and if glucose tolerance test may be useful as a diagnostic tool by predicting potential improvement of insulin sensitivity after biochemical cure of pHPT.

DETAILED DESCRIPTION:
To be conducted at the Karolinska University Hospital, Stockholm. Patients with fb-glucos >6.1 and HbA1c without medical treatment will be included after informed consent and randomised to parathyroidectomy (PTX) within three months or not. The groups will be examined 4 ±4 weeks before and 12±2 weeks after PTX, similar for the control group. The number of participants will be estimated by power calculations based on a pilot study including 20 patients.

The test protocol includes glucose load with control of glucose and insulin, (0, 30, 60 and 120 min) together with measurement of markers of oxidative stress and inflammation.

ELIGIBILITY:
Inclusion Criteria:

* primary hyperparathyroidism and fb-glukos>6,1 and/or HbA1c > 39 mmol/mol

Exclusion Criteria:

* Treatment with insulin, sulfonylurea or metformin

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-10; Primary Completion 2021-12 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
glucose tolerance test with estimation of insulin resistance | 3 months
  Homa IR
quality of life - self estimation protocol | 3 months
  EORTC QLQ-C30

SECONDARY OUTCOMES:
psychological wellbeing | 3 months
  POMS
anxiety, depression | 6 months
  HAD
cognition | 6 months
  MoCA-Test

CONTACTS AND LOCATIONS:
Overall Officials: Inga-Lena Nilsson, MD, PhD, Principal Investigator — Karolinska University Hospital
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Norenstedt S, Pernow Y, Brismar K, Saaf M, Ekip A, Granath F, Zedenius J, Nilsson IL. Primary hyperparathyroidism and metabolic risk factors, impact of parathyroidectomy and vitamin D supplementation, and results of a randomized double-blind study. Eur J Endocrinol. 2013 Oct 21;169(6):795-804. doi: 10.1530/EJE-13-0547. Print 2013 Dec. PMID 24026893
- See also: Regional program — http://www.viss.nu/Handlaggning/Vardprogram/Endokrina-organ/Prediabetes/